CLINICAL TRIAL: NCT01851330
Title: A Phase 3, Multicenter, Randomized, Open-Label Study to Investigate the Efficacy and Safety of Sofosbuvir/Ledipasvir Fixed-Dose Combination ± Ribavirin for 8 Weeks and Sofosbuvir/Ledipasvir Fixed-Dose Combination for 12 Weeks in Treatment-Naive Subjects With Chronic Genotype 1 HCV Infection
Brief Title: Safety and Efficacy of Ledipasvir/Sofosbuvir Fixed-Dose Combination ± Ribavirin for the Treatment of HCV (ION-3)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-337-0108
Record Dates: First submitted 2013-05-03; First posted 2013-05-10 (Estimated); Results first posted 2014-12-30 (Estimated); Last update posted 2018-11-16 (Actual); Status verified 2014-12

CONDITIONS: Chronic Hepatitis C Virus
Keywords: HCV genotype 1 (GT-1); HCV; Sustained Virologic Response; Direct Acting Antiviral; Combination Therapy; GS-7977; GS-5885; Ribavirin; Open Label; Sofosbuvir; Additional relevant MeSH terms:; Hepatitis; Hepatitis, Chronic; Hepatitis C; Hepatitis C, Chronic; Liver Diseases; Digestive System Diseases; Hepatitis, Viral, Human; Virus Diseases; Enterovirus Infections; Picornaviridae Infections; RNA Virus Infections; Flaviviridae Infections; Antiviral Agents; Anti-Infective Agents; Therapeutic Uses; Pharmacologic Actions; Antimetabolites; Molecular Mechanisms of Pharmacological Action
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis; Hepatitis, Chronic; Hepatitis C; Liver Diseases; Digestive System Diseases; Hepatitis, Viral, Human; Virus Diseases; Enterovirus Infections; Picornaviridae Infections; RNA Virus Infections; Flaviviridae Infections | interventions — ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- LDV/SOF 8 Week (Experimental): Participants will receive LDV/SOF FDC for 8 weeks.
  Interventions: Drug: LDV/SOF
- LDV/SOF+RBV 8 Week (Experimental): Participants will receive LDV/SOF FDC plus RBV for 8 weeks.
  Interventions: Drug: LDV/SOF; Drug: RBV
- LDV/SOF 12 Week (Experimental): Participants will receive LDV/SOF FDC for 12 weeks.
  Interventions: Drug: LDV/SOF

INTERVENTIONS:
Drug: LDV/SOF — LDV 90 mg/SOF 400 mg FDC tablet administered orally once daily
  Other Names: Harvoni®; GS-5885/GS-7977
Drug: RBV — Ribavirin (RBV) tablets administered orally in a divided daily dose according to package insert weight-based dosing recommendations (< 75 kg = 1000 mg and ≥ 75 kg = 1200 mg)
  Arms: LDV/SOF+RBV 8 Week

SUMMARY:
This study is to evaluate the safety, tolerability, and antiviral efficacy of ledipasvir/sofosbuvir (LDV/SOF) fixed-dose combination (FDC) with or without ribavirin (RBV) administered for 8 or 12 weeks in treatment-naive participants with chronic genotype 1 HCV infection.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18, with chronic genotype 1 HCV infection
* HCV treatment-naive
* HCV RNA > 10,000 IU/mL at screening
* Screening laboratory values within defined thresholds
* Use of two effective contraception methods if female of childbearing potential or sexually active male

Exclusion Criteria:

* Pregnant or nursing female or male with pregnant female partner
* Presence of cirrhosis
* Coinfection with HIV or hepatitis B virus (HBV)
* Current or prior history of clinical hepatic decompensation
* Chronic use of systemic immunosuppressive agents
* History of clinically significant illness or any other medical disorder that may interfere with subject treatment, assessment or compliance with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 647 (Actual)
Dates: Start 2013-05; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert H. Hyland, DPhil, Study Director — Gilead Sciences
Locations (52):
- United States (52):
  - Birmingham, Alabama
  - La Jolla, California
  - Los Angeles, California
  - Palo Alto, California
  - Sacramento, California
  - San Diego, California
  - San Francisco, California
  - Aurora, Colorado
  - Englewood, Colorado
  - Washington D.C., District of Columbia
  - Gainesville, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Orlando, Florida
  - Wellington, Florida
  - Atlanta, Georgia
  - Decatur, Georgia
  - Marietta, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Bowling Green, Kentucky
  - Baton Rouge, Louisiana
  - Baltimore, Maryland
  - Lutherville, Maryland
  - Boston, Massachusetts
  - Novi, Michigan
  - Kansas City, Missouri
  - St Louis, Missouri
  - Albuquerque, New Jersey
  - Berlin, New Jersey
  - Hillsborough, New Jersey
  - Santa Fe, New Mexico
  - Binghamton, New York
  - Manhasset, New York
  - New York, New York
  - Chapel Hill, North Carolina
  - Fayetteville, North Carolina
  - Statesville, North Carolina
  - Winston-Salem, North Carolina
  - Philadelphia, Pennsylvania
  - Providence, Rhode Island
  - Germantown, Tennessee
  - Nashville, Tennessee
  - Arlington, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Fairfax, Virginia
  - Falls Church, Virginia
  - Newport News, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
  - Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

REFERENCES:
- [Derived] Grebely J, Mauss S, Brown A, Bronowicki JP, Puoti M, Wyles D, Natha M, Zhu Y, Yang J, Kreter B, Brainard DM, Yun C, Carr V, Dore GJ. Efficacy and Safety of Ledipasvir/Sofosbuvir With and Without Ribavirin in Patients With Chronic HCV Genotype 1 Infection Receiving Opioid Substitution Therapy: Analysis of Phase 3 ION Trials. Clin Infect Dis. 2016 Dec 1;63(11):1405-1411. doi: 10.1093/cid/ciw580. Epub 2016 Aug 23. PMID 27553375
- [Derived] Kowdley KV, Gordon SC, Reddy KR, Rossaro L, Bernstein DE, Lawitz E, Shiffman ML, Schiff E, Ghalib R, Ryan M, Rustgi V, Chojkier M, Herring R, Di Bisceglie AM, Pockros PJ, Subramanian GM, An D, Svarovskaia E, Hyland RH, Pang PS, Symonds WT, McHutchison JG, Muir AJ, Pound D, Fried MW; ION-3 Investigators. Ledipasvir and sofosbuvir for 8 or 12 weeks for chronic HCV without cirrhosis. N Engl J Med. 2014 May 15;370(20):1879-88. doi: 10.1056/NEJMoa1402355. Epub 2014 Apr 10. PMID 24720702

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at a total of 59 study sites in the United States. The first participant was screened on 06 May 2013. The last participant observation occurred on 07 March 2014.
Pre-assignment Details: 831 participants were screened.
Groups:
- LDV/SOF 8 Week: Ledipasvir (LDV) 90 mg/sofosbuvir (SOF) 400 mg fixed-dose combination (FDC) tablet once daily for 8 weeks
- LDV/SOF+RBV 8 Week: LDV 90 mg/SOF 400 mg FDC tablet once daily plus ribavirin (RBV) tablets (1000 or 1200 mg daily based on weight) for 8 weeks
- LDV/SOF 12 Week: LDV 90 mg/SOF 400 mg FDC tablet once daily for 12 weeks
Period: Overall Study
Arm/Group | LDV/SOF 8 Week | LDV/SOF+RBV 8 Week | LDV/SOF 12 Week
Started | 215 | 216 | 216
Completed | 202 | 200 | 204
Not Completed | 13 | 16 | 12
Not completed — Lack of Efficacy | 10 | 9 | 2
Not completed — Lost to Follow-up | 1 | 6 | 9
Not completed — Withdrew Consent | 2 | 1 | 0
Not completed — Investigator's Discretion | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants were randomized and received at least one dose of study medication.
Groups:
- LDV/SOF 8 Week: LDV 90 mg/SOF 400 mg FDC tablet once daily for 8 weeks
- LDV/SOF+RBV 8 Week: LDV 90 mg/SOF 400 mg FDC tablet once daily plus RBV tablets (1000 or 1200 mg daily based on weight) for 8 weeks
- Total: Total of all reporting groups
Arm/Group | LDV/SOF 8 Week | LDV/SOF+RBV 8 Week | LDV/SOF 12 Week | Total
Number analyzed (Participants) | 215 | 216 | 216 | 647
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (10.2) | 51 (11.7) | 53 (10.6) | 52 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender was collected as "Sex at Birth."
  Participants
    Female | 85 | 99 | 88 | 272
    Male | 130 | 117 | 128 | 375
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 45 | 36 | 42 | 123
  White | 164 | 176 | 167 | 507
  Asian | 5 | 2 | 3 | 10
  American Indian/Alaska Native | 0 | 1 | 0 | 1
  Hawaiian or Pacific Islander | 0 | 1 | 0 | 1
  Other | 1 | 0 | 3 | 4
  Not Disclosed | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 13 | 12 | 14 | 39
  Not Hispanic or Latino | 200 | 204 | 202 | 606
  Not Disclosed | 2 | 0 | 0 | 2
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.5 (0.76) | 6.4 (0.69) | 6.4 (0.76) | 6.5 (0.74)
HCV RNA Category [Number; unit: participants]
  < 800,000 IU/mL | 34 | 45 | 44 | 123
  ≥ 800,000 IU/mL | 181 | 171 | 172 | 524
HCV Genotype [Number; unit: participants]
  Genotype 1 (no confirmed subtype) | 1 | 0 | 0 | 1
  Genotype 1a | 171 | 172 | 172 | 515
  Genotype 1b | 43 | 44 | 44 | 131
IL28b Status [Number; unit: participants] — CC, CT, and TT alleles are different forms of the IL28b gene.
  participants
    CC | 56 | 60 | 56 | 172
    CT | 120 | 128 | 124 | 372
    TT | 39 | 28 | 36 | 103

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, 25 IU/mL) 12 weeks following the last dose of study drug.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set: participants were randomized and received at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF 8 Week | LDV/SOF+RBV 8 Week | LDV/SOF 12 Week
Number analyzed (Participants) | 215 | 216 | 216
percentage of participants | 94.0 | 93.1 | 96.3
Statistical Analysis 1: Comparison: LDV/SOF 8 Week; Test type: Superiority or Other; p < 0.001, Binomial test — The p-value for the comparison of the LDV/SOF 8 week group against the adjusted historical null rate (60%) was based on a 2-sided 1-sample binomial test
Statistical Analysis 2: Comparison: LDV/SOF+RBV 8 Week; Test type: Superiority or Other; p < 0.001, Binomial test — The p-value for the comparison of the LDV/SOF+RBV 8 week group against the adjusted historical null rate (60%) was based on a 2-sided 1-sample binomial test
Statistical Analysis 3: Comparison: LDV/SOF 12 Week; Test type: Superiority or Other; p < 0.001, Binomial test — The p-value for the comparison of the LDV/SOF 12 week group against the adjusted historical null rate (60%) was based on a 2-sided 1-sample binomial test
Statistical Analysis 4: Comparison: LDV/SOF+RBV 8 Week vs LDV/SOF 12 Week; Test type: Non-Inferiority or Equivalence — Noninferiority would be demonstrated if the lower bound of the confidence interval (CI) for the difference between groups was greater than -12%; Difference in proportions = -3.2, 97.5% CI 2-sided [-8.3 to 1.8] — Difference in proportions between treatment groups and associated confidence interval (CI) were calculated based on stratum-adjusted Mantel-Haenszel proportions
Statistical Analysis 5: Comparison: LDV/SOF 8 Week vs LDV/SOF 12 Week; Test type: Non-Inferiority or Equivalence — Noninferiority would be demonstrated if the lower bound of the CI for the difference between groups was greater than -12%; Difference in proportions = -2.3, 97.5% CI 2-sided [-7.2 to 2.5] — [estimate comment as in outcome 1, analysis 4]
Statistical Analysis 6: Comparison: LDV/SOF 8 Week vs LDV/SOF+RBV 8 Week; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 5]; Difference in proportions = 0.9, 95% CI 2-sided [-3.9 to 5.7] — [estimate comment as in outcome 1, analysis 4]

2. Primary Outcome: Incidence of Adverse Events Leading to Permanent Discontinuation From Any Study Drug
Description: The percentage of participants who experienced an adverse event leading to permanent discontinuation from any study drug was summarized.
Time Frame: Up to 12 weeks
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF 8 Week | LDV/SOF+RBV 8 Week | LDV/SOF 12 Week
Number analyzed (Participants) | 215 | 216 | 216
percentage of participants | 0 | 0.9 | 0.9

3. Secondary Outcome: Percentage of Participants With Sustained Virologic Response at 4 and 24 Weeks After Discontinuation of Therapy (SVR4 and SVR24)
Description: SVR4 and SVR24 were defined as HCV RNA < LLOQ at 4 and 24 weeks following the last dose of study drug, respectively.
Time Frame: Posttreatment Weeks 4 and 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF 8 Week | LDV/SOF+RBV 8 Week | LDV/SOF 12 Week
Number analyzed (Participants) | 215 | 216 | 216
percentage of participants
  SVR4 | 96.3 | 94.9 | 96.3
  SVR24 | 94.0 | 93.1 | 96.3

4. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 2
Time Frame: Week 2
Population: Participants in the Full Analysis Set with Available Data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF 8 Week | LDV/SOF+RBV 8 Week | LDV/SOF 12 Week
Number analyzed (Participants) | 215 | 214 | 216
percentage of participants | 88.4 | 91.1 | 91.2

5. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 4
Time Frame: Week 4
Population: Participants in the Full Analysis Set with Available Data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF 8 Week | LDV/SOF+RBV 8 Week | LDV/SOF 12 Week
Number analyzed (Participants) | 216 | 213 | 216
percentage of participants | 100.0 | 99.1 | 100.0

6. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 8
Time Frame: Week 8
Population: Participants in the Full Analysis Set with Available Data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF 8 Week | LDV/SOF+RBV 8 Week | LDV/SOF 12 Week
Number analyzed (Participants) | 215 | 213 | 214
percentage of participants | 100.0 | 100.0 | 99.5

7. Secondary Outcome: Change From Baseline in HCV RNA at Week 2
Time Frame: Baseline; Week 2
Population: Participants in the Full Analysis Set with Available Data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | LDV/SOF 8 Week | LDV/SOF+RBV 8 Week | LDV/SOF 12 Week
Number analyzed (Participants) | 215 | 212 | 212
log10 IU/mL | -5.06 (0.752) | -5.01 (0.675) | -4.99 (0.750)

8. Secondary Outcome: Change From Baseline in HCV RNA at Week 4
Time Frame: Baseline; Week 4
Population: Participants in the Full Analysis Set with Available Data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | LDV/SOF 8 Week | LDV/SOF+RBV 8 Week | LDV/SOF 12 Week
Number analyzed (Participants) | 215 | 212 | 216
log10 IU/mL | -5.12 (0.760) | -5.05 (0.682) | -5.05 (0.758)

9. Secondary Outcome: Change From Baseline in HCV RNA at Week 8
Time Frame: Baseline; Week 8
Population: Participants in the Full Analysis Set with Available Data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | LDV/SOF 8 Week | LDV/SOF+RBV 8 Week | LDV/SOF 12 Week
Number analyzed (Participants) | 215 | 213 | 213
log10 IU/mL | -5.12 (0.760) | -5.05 (0.683) | -5.04 (0.761)

10. Secondary Outcome: Percentage of Participants Experiencing Virologic Failure
Description: Virologic failure was defined as on-treatment virologic failure or virologic relapse.
  * On-Treatment Virologic Failure was defined as
    * Breakthrough (confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while on treatment), or
    * Rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment), or
    * Non-response (HCV RNA persistently ≥ LLOQ through 8 weeks of treatment) Virologic relapse was defined as confirmed HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at last on-treatment visit.
Time Frame: Baseline to posttreatment Week 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF 8 Week | LDV/SOF+RBV 8 Week | LDV/SOF 12 Week
Number analyzed (Participants) | 215 | 216 | 216
percentage of participants
  On-treatment virologic failure | 0 | 0 | 0
  Virologic relapse | 5.1 | 4.2 | 1.4

ADVERSE EVENTS:
Time Frame: Up to 12 weeks plus 30 days
Description: Safety Analysis Set
Arm/Group | LDV/SOF 8 Week | LDV/SOF+RBV 8 Week | LDV/SOF 12 Week
Serious Adverse Events (participants affected / at risk) | 4/215 | 1/216 | 5/216
Other Adverse Events (participants affected / at risk) | 146/215 | 166/216 | 150/216
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LDV/SOF 8 Week (N=215) | LDV/SOF+RBV 8 Week (N=216) | LDV/SOF 12 Week (N=216)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 0 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 1
Haemothorax 0 (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LDV/SOF 8 Week (N=215) | LDV/SOF+RBV 8 Week (N=216) | LDV/SOF 12 Week (N=216)
Anaemia (Blood and lymphatic system disorders) | 2 | 17 | 2
Nausea (Gastrointestinal disorders) | 15 | 39 | 24
Diarrhoea (Gastrointestinal disorders) | 15 | 13 | 9
Constipation (Gastrointestinal disorders) | 9 | 12 | 8
Fatigue (General disorders) | 45 | 75 | 49
Irritability (General disorders) | 3 | 29 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 12 | 16
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 12 | 6
Headache (Nervous system disorders) | 30 | 54 | 33
Dizziness (Nervous system disorders) | 6 | 13 | 9
Insomnia (Psychiatric disorders) | 11 | 26 | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 12 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 11 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 20 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 16 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years